CLINICAL TRIAL: NCT01007487
Title: Wound Retractor or Protector? Efficacy of a Plastic Wound Retractor (Alexis®) in Impeding Translocation of Enteric Bacteria to the Surgical Incision Site in Abdominal Surgery.
Brief Title: Plastic Wound Retractors and Bacterial Translocation in Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Desmond Winter, St Vincent's University Hospital, Ireland
Other Study IDs: HMSVUH1
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2009-11

CONDITIONS: Bacterial Translocation; Surgical Site Infection; Abdominal Surgery; Wound Infection
Keywords: Plastic wound protector; Plastic wound retractor; Bacterial translocation; Surgical site infection; Abdominal surgery; Wound infection
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: Plastic wound retractors reduce passage of bacteria from the abdomen to the surgical incision site in abdominal surgery

Currently, plastic wound retractors are used in abdominal surgery to facilitate access to the abdominal cavity. This study aims to establish whether they also prevent bacteria crossing from the abdominal cavity to the surgical incision site. Patients undergoing abdominal surgery in which a plastic wound retractor (Alexis®)is used are eligible for inclusion in the study. Swabs are taken from the inside and the outside of the plastic wound retractor prior to removing the retractor from the abdomen. The bacterial flora from swabs taken inside and outside the plastic wound protector are then compared to see if there is any difference between inside and outside the retractor. Bacteria are classified as 'enteric'(i.e. from the gastrointestinal tract) or 'skin' bacteria, depending on their usual location. The study aims to establish whether a plastic wound retractor (Alexis®) reduces translocation of enteric bacteria to the surgical incision site.

DETAILED DESCRIPTION:
Plastic wound retractors are currently used in abdominal surgery for wound retraction. They allow access to intra-abdominal organs through an incision in abdominal surgery. Plastic wound retractors may also act as a barrier to bacterial translocation from the abdominal cavity to the wound. The purpose of this study was to compare microbial flora from inside and outside the plastic wound retractor to establish whether plastic wound retractors affect bacterial translocation.

METHODS This multi-centre prospective observational study is being conducted between November 2007 and January 2010. Patients undergoing elective or emergency abdominal surgery in which an Alexis® wound retractor is used are eligible for inclusion in the study. Swabs are taken from inside and outside the Alexis® wound protector immediately prior to removal of the wound protector from the abdominal cavity. Swabs undergo gram stain and culture. "Inside" the wound swab is defined as the part of the wound protector in contact with the intra-abdominal organs, "outside" is the part in contact with the skin and subcutaneous tissues. Results from inside and outside swabs are then compared to establish whether there is a difference in bacterial flora. The study aims to establish whether a plastic wound retractor (Alexis®) reduces translocation of enteric bacteria to the surgical incision site.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing abdominal surgery in which a plastic wound retractor is used

Exclusion Criteria:

* N/A

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing abdominal surgery in which a plastic wound retractor is used.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Comparison of inside swabs positive for enteric bacteria and outside swabs positive for enteric bacteria. | 2 years

SECONDARY OUTCOMES:
Comparison of bacteria isolated from intraoperative swabs and subsequent post-operative swabs (<30days post-operatively) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Winter, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (2):
- Ireland (2):
  - Mater Misericordiae University Hospital, Eccles Street, Dublin
  - St. Vincent's University Hospital, Elm Park, Dublin